CLINICAL TRIAL: NCT02138617
Title: Genotype-Directed Phase II Study Of Higher Dose Of Irinotecan In First-Line Metastatic Colorectal Cancer Patients Treated With Folfiri Plus Bevacizumab
Brief Title: Genotype-Directed Study Of Irinotecan Dosing In FOLFIRI + BevacizumabTreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1317
Record Dates: First submitted 2014-05-01; First posted 2014-05-14 (Estimated); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
Keywords: Colon Cancer; Irinotecan; FOLFIRI; Genotyping; UGT1A1
MeSH Terms: conditions — Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- *1/*1 Genotype (Experimental): FOLFIRI (5-fluorouracil (5-FU), leucovorin, irinotecan) Irinotecan dose 310 mg/m2,(IV, Day 1, 15); Bevacizumab (IV, Day 1, 15), repeat treatment cycle every 28 days.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab
- *1/*28 Genotype (Experimental): FOLFIRI (5-fluorouracil (5-FU), leucovorin, irinotecan) Irinotecan dose 260 mg/m2, FOLFIRI (IV, Day 1, 15); Bevacizumab (IV, Day 1, 15), repeat treatment cycle every 28 days.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab
- *28/*28 (Experimental): FOLFIRI (5-fluorouracil (5-FU), leucovorin, irinotecan) Irinotecan dose 180 mg/m2, FOLFIRI (IV, Day 1, 15); Bevacizumab (IV, Day 1, 15), repeat treatment cycle every 28 days.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: 5-Fluorouracil — 400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hours, Day 1 and Day 15 .
  Other Names: 5-FU; Adrucil
Drug: Leucovorin — 200-400 mg/m2 IV over 2 hours, Day 1 and Day 15
  Other Names: LV; leucovorin calcium; folinic acid; citrovorum factor
Drug: Irinotecan — IV infusion over 90 minutes, dosed at 180, 260 or 310 mg/m2 based on genotype.
  Other Names: Camptosar; Novaplus Irinotecan Hydrochloride
Drug: Bevacizumab — Bevacizumab (5 mg/kg IV infused as per institutional policy, IV, Day 1, 15)
  Other Names: Avastin; MVASI

SUMMARY:
This study involves standard combination chemotherapy treatment for colon cancer, 5-Fluorouracil (5FU), leucovorin and irinotecan (known as FOLFIRI), plus bevacizumab (Avastin). The study is designed to test the FOLFIRI regimen based on certain characteristics of a person's genetic makeup or "genes". Genes are made of DNA and determine not only inherited traits or appearance (hair and eye color, height, body type, etc.) but also play an important role in health and how the body responds to illness and treatments for those illnesses.

In this study, the investigators will examine the relationship between a patient's genes (DNA), or "genotype", and how the patient's body breaks down and removes or "metabolizes" the anti-cancer drug irinotecan. Circulating blood level of irinotecan plays an important role in how well this drug works against a patient's cancer as well as the adverse side effects the patient may experience. The current standard dose of irinotecan was determined in clinical trials without knowing individual genotypes and thus does not take into account a patient's ability to metabolize irinotecan. This means that based on one genotype the current standard dose of irinotecan may be correct or based on other genotypes the standard dose could result in lower and possibly less effective blood levels and result in significant under-dosing of irinotecan.

Based on genotype the patient will be assigned to one of the following doses of irinotecan:

* 180 mg/m2 (standard dose)
* 260 mg/m2
* 310 mg/m2

The purpose of this research study is to determine if dosing irinotecan based on genotype is effective and safe for patients with colon cancer. Patient genotype will be determined from a small sample of blood and a laboratory test or "assay" performed at University of North Carolina Laboratories. For the purpose of this study, this assay is new and considered to be "investigational". This means that the genotype assay used in this study has not yet been approved by the FDA for determining irinotecan dose levels in patients with colon cancer.

DETAILED DESCRIPTION:
This phase II multicenter clinical trial will use a genotype-guided dosing strategy for irinotecan to prospectively analyze efficacy in 100 metastatic colorectal cancer patients (mCRC) receiving FOLFIRI (5-fluorouracil (5-FU), leucovorin, irinotecan) plus bevacizumab. Irinotecan is detoxified and excreted primarily by glucuronidation in the liver via the isoenzyme uridine diphosphate glucuronosyl transferase (UGT1A1). Common variants in UGT1A1 alter the rate of glucuronidation and thus alter exposure to irinotecan.

The UGT1A1 *28 allele results in slower irinotecan glucuronidation, and thus greater exposure to its active metabolite SN-38. At the standard irinotecan dose used in FOLFIRI (180 mg/m2; established prior to our understanding of the importance of genotype in the rate of this drug's metabolism), there is a small increased risk of neutropenia in *28 homozygotes. However, the risk of clinically important consequences of neutropenia, such as febrile neutropenia and infection, are not significantly increased. Patients with other genotypes have a quite low risk of adverse effects suggesting patients with these low risk genotypes may tolerate higher doses of irinotecan in FOLFIRI. This finding was demonstrated in a phase I study in which *1/*28 and *1/*1 genotypes were able to tolerate escalating doses of irinotecan up to 260 mg/m2 and 310 mg/m2, respectively.

The central hypothesis of this trial is that increasing the irinotecan dose in *1/*28 and *1/*1 genotypes will increase the overall benefit of FOLFIRI for patients with mCRC as these two groups are likely under-dosed with the current dosing regimen. Eligible patients will be genotyped for UGT1A1 and assigned into 1 of 3 different dosing groups, based on their relative rate of metabolism. The primary objective of this trial is to estimate progression-free survival (PFS), and secondary objectives include characterization of toxicity and objective response rate (OR; complete response (CR) + partial response (PR)).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to participate in this study:

1. An Institutional Review Board-approved informed consent obtained and signed
2. Age ≥ 18 years
3. Histological or cytological documentation of adenocarcinoma of the colon or rectum
4. Measurable or non-measurable (but evaluable) disease as defined via RECIST 1.1
5. Metastatic disease not amenable to surgical resection with curative intent
6. No prior chemotherapy for metastatic disease
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see section 11.1, Appendix A)
8. Adequate bone marrow, renal and hepatic function, as evidenced by the following:

   * absolute neutrophil count (ANC) ≥1,500/mm3
   * platelets ≥100,000/mm3
   * hemoglobin ≥9.0 g/dL
   * serum creatinine ≤1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤3x ULN ( ≤5.0 × ULN for patients with liver involvement of their cancer
   * Bilirubin ≤1.5 X ULN
   * Alkaline phosphatase ≤3 x ULN (≤5 x ULN with liver involvement of their cancer)
9. Willing to undergo UGT1A1 genotyping
10. Negative pregnancy test (urine or serum), within 7 day prior to Day 1 of FOLFIRI in women of childbearing potential
11. Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.

Exclusion Criteria

1. UGT1A1 genotype other than *1/*1, *1/*28, or *28/*28
2. Known dihydropyrimidine dehydrogenase (DPD) deficiency
3. Prior treatment with irinotecan and/or bevacizumab
4. Unable or unwilling to discontinue (and substitute if necessary) use of prohibited drugs for at least 14 days (fruits and juices for at least 7 days) prior to Day 1 of FOLFIRI + bevacizumab initiation (see section 11.2, Appendix B, for list of prohibited drugs)
5. Inadequately controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg)
6. Prior history of hypertensive encephalopathy
7. Active cardiac disease including any of the following:

   * New York Heart Association (NYHA) Grade II or greater congestive heart failure (see section 11.3, Appendix C)
   * History of myocardial infarction or unstable angina within 6 months prior to Day 1
   * History of stroke or transient ischemic attack within 6 months prior to Day 1 of FOLFIRI + bevacizumab initiation
8. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of FOLFIRI + bevacizumab initiation
9. History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1 of FOLFIRI + bevacizumab initiation
10. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of FOLFIRI + bevacizumab initiation or anticipation of need for major surgical procedure during the course of the study
12. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1 of FOLFIRI + bevacizumab initiation
13. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1 of FOLFIRI + bevacizumab initiation
14. Serious, non-healing wound, active ulcer, or untreated bone fracture
15. Proteinuria as demonstrated by:

    Urine protein: creatinine (UPC) ratio ≥ 1.0 at screening OR Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
16. Any serious uncontrolled medical disorder that would impair the ability of the subject to receive protocol-driven therapy
17. Other anti-cancer or investigational therapy while patients are on study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sannoff, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (7):
- United States (7):
  - IU Simon Cancer Center, Indianapolis, Indiana
  - IU Arnett Hospital, Lafayette, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Healthcare Systems, Charlotte, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Bon Secours Cancer Institute, Midlothian, Virginia

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://cancer.unc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in the study between 5/6/2014 and 08/29/20192 at eight cancer centers in the United States.
Period: Overall Study
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
Started | 47 | 43 | 10
Completed | 0 | 0 | 0
Not Completed | 47 | 43 | 10
Not completed — Death | 1 | 2 | 2
Not completed — Adverse Event | 8 | 5 | 2
Not completed — Disease Progression | 20 | 13 | 4
Not completed — Withdrawal by Subject | 7 | 10 | 2
Not completed — other complicating disease | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 7 | 6 | 0
Not completed — financial reason | 0 | 1 | 0
Not completed — other therapy | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28 | Total
Number analyzed (Participants) | 47 | 43 | 10 | 100
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 79] | 59 [19 to 72] | 62 [52 to 76] | 59 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 8 | 48
  Male | 25 | 25 | 2 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 41 | 43 | 10 | 94
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 2 | 12
  White | 40 | 35 | 8 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 43 | 10 | 100

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free Free Survival is defined as the time from day 1 (D1) of treatment to progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST)1.1 or death from any cause. Radiographic response will be measured by RECIST, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of registration until date of first documented progression up to 8 years.
Population: Participants started the study and response assessments were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
Number analyzed (Participants) | 41 | 36 | 6
Participants
  The response was achieved, or the disease remained stable | 38 | 34 | 6
  Disease Progression | 3 | 2 | 0

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: The toxicity profile when irinotecan is dosed according to isoenzyme uridine diphosphate glucuronosyl transferase (UGT1A1) Genotypes was evaluated and Grade 3 or higher adverse events were reported. Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).
Time Frame: From date of registration up to 8 years.
Population: Participants started the study and adverse event assessments were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
Number analyzed (Participants) | 47 | 39 | 10
Participants
  General Fatigue | 2 | 5 | 1
  Febrile neutropenia | 1 | 0 | 1
  Neutropenia | 24 | 20 | 5
  Sepsis | 1 | 0 | 1
  Leukopenia | 2 | 3 | 3
  Lymphopenia | 0 | 5 | 1
  Anemia | 1 | 3 | 3
  Thrombocytopenia | 2 | 2 | 3
  Nausea | 1 | 2 | 1
  Vomiting | 2 | 3 | 1
  Diarrhea | 6 | 5 | 1
  Mucositis | 4 | 3 | 2
  Hypertension | 5 | 4 | 1

3. Secondary Outcome: Overall Response
Description: Overall Response (OR =Complete Response +Partial Response) will be defined per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 years
Population: Participants started the study and response assessments were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
Number analyzed (Participants) | 41 | 36 | 6
Participants
  Complete Response or Partial Response was achieved | 28 | 20 | 3
  Stable disease or progression | 13 | 16 | 3

4. Secondary Outcome: Overall Survival Rate
Description: The Overall Survival rate (OS) is defined as the percentage of participants alive after time from D1 of treatment to death from any cause.
Time Frame: 8 years
Population: Participants started the study.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
Number analyzed (Participants) | 43 | 39 | 9
months | 26.5 [19.1 to 32.9] | 25.9 [17.6 to 37.7] | 13.4 [2.3 to 20.5]

ADVERSE EVENTS:
Time Frame: Up to 8 years.
Description: Adverse events were collected from day one of the study treatment. Per protocol, all hospitalizations were graded as serious adverse events.
Arm/Group | *1/*1 Genotype | *1/*28 Genotype | *28/*28
All-Cause Mortality (participants affected / at risk) | 38/47 | 34/43 | 9/10
Serious Adverse Events (participants affected / at risk) | 14/47 | 13/43 | 4/10
Other Adverse Events (participants affected / at risk) | 47/47 | 43/43 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | *1/*1 Genotype (N=47) | *1/*28 Genotype (N=43) | *28/*28 (N=10)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 0
colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 1
colonic perforation (Gastrointestinal disorders) | 1 | 2 | 1
colonic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Urostomy leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1
White blood cell decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 3 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | *1/*1 Genotype (N=47) | *1/*28 Genotype (N=43) | *28/*28 (N=10)
Anemia (Blood and lymphatic system disorders) | 28 | 25 | 8
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 2 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Blurred vision (Eye disorders) | 4 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 | 0
Floaters (Eye disorders) | 1 | 1 | 1
Watering eyes (Eye disorders) | 4 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 15 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Anal mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colonic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 23 | 2
Diarrhea (Gastrointestinal disorders) | 30 | 31 | 6
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 4 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 3 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 4 | 4 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 29 | 23 | 4
Nausea (Gastrointestinal disorders) | 32 | 35 | 7
Oral dysesthesia (Gastrointestinal disorders) | 0 | 2 | 0
Oral hemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 3 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 17 | 20 | 6
Chills (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 8 | 5 | 1
Fatigue (General disorders) | 30 | 29 | 6
Fever (General disorders) | 3 | 5 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 2 | 0
Infusion related reaction (General disorders) | 2 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 8 | 7 | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0
Cecal infection (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Gum infection (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 3 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 3 | 1
Mucosal infection (Infections and infestations) | 2 | 0 | 2
Nail infection (Infections and infestations) | 2 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Penile infection (Infections and infestations) | 1 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Upper respiratory infection (Infections and infestations) | 7 | 2 | 1
Urinary tract infection (Infections and infestations) | 7 | 3 | 1
Bruising (Injury, poisoning and procedural complications) | 5 | 5 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 13 | 4 | 0
Alkaline phosphatase increased (Investigations) | 15 | 13 | 1
Aspartate aminotransferase increased (Investigations) | 16 | 10 | 1
Blood bilirubin increased (Investigations) | 3 | 2 | 4
Cholesterol high (Investigations) | 1 | 0 | 0
Creatine Phosphokinase increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 8 | 10 | 1
INR (international normalized ratio) (Investigations) | 1 | 0 | 0
Investigations - Other, specify (Investigations) | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 11 | 14 | 3
Neutrophil count decreased (Investigations) | 37 | 31 | 7
Platelet count decreased (Investigations) | 12 | 12 | 5
Weight gain (Investigations) | 1 | 1 | 0
Weight loss (Investigations) | 8 | 7 | 4
White blood cell decreased (Investigations) | 21 | 18 | 5
Anorexia (Metabolism and nutrition disorders) | 26 | 22 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 8 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 5 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 7 | 9 | 2
Hypernatremia (Metabolism and nutrition disorders) | 2 | 4 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 17 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 9 | 3
Hypokalemia (Metabolism and nutrition disorders) | 20 | 17 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 14 | 2
Hyponatremia (Metabolism and nutrition disorders) | 12 | 11 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 6 | 1
Dysgeusia (Nervous system disorders) | 4 | 5 | 0
Headache (Nervous system disorders) | 16 | 9 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 4 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 3 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 2 | 3 | 1
Insomnia (Psychiatric disorders) | 15 | 14 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 6 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 14 | 14 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Reproductive system and breast disorders) | 2 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1 | 0
Urine discoloration (Renal and urinary disorders) | 2 | 0 | 0
Erectile dysfunction (Renal and urinary disorders) | 1 | 2 | 1
Genital edema (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 13 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 4 | 3 | 0
Hypertension (Vascular disorders) | 18 | 15 | 4
Hypotension (Vascular disorders) | 0 | 2 | 2
Thromboembolic event (Vascular disorders) | 6 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subcontractor agrees that the first publication of the Study results will be made by Institution as a multi-site publication. Subcontractor can publish its site-specific results after Institution's publication, 12 months post-study completion, or upon Institution's notice. Subcontractor must provide Institution 30 days for manuscript review and may delay publication for 45 days for patent filing. Institution will register the Study and post results as required by law.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT02138617/Prot_SAP_000.pdf